CLINICAL TRIAL: NCT04499313
Title: The Outcome of Dexamethasone and Methylprednisolone Treatment for Patients With ARDS Caused by COVID-19
Brief Title: Dexamethasone Vs Methylprednisolone for the Treatment of Patients With ARDS Caused by COVID-19
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chattogram General Hospital (Other Government)
Collaborators: Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10000753
Record Dates: First submitted 2020-07-27; First posted 2020-08-05 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Covid19; ARDS
Keywords: COVID 19; Dexamethasone; Methylprednisolone; ARDS
MeSH Terms: conditions — COVID-19 | interventions — Dexamethasone; Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A: Dexamethasone (Active Comparator): Dexamethasone (20 mg/iv/daily/from Day 1 of randomization, followed by a tapering dose according to the patient's condition.
  Interventions: Drug: Dexamethasone
- Group B: Methylprednisolone (Active Comparator): Methylprednisolone Sodium Succinate at a dose of 0.5mg/kg (Injectable solution)
  Interventions: Drug: Methylprednisolone

INTERVENTIONS:
Drug: Dexamethasone — Injectable solution
  Arms: Group A: Dexamethasone
Drug: Methylprednisolone — Injectable solution
  Arms: Group B: Methylprednisolone

SUMMARY:
A randomized clinical trial designed and intended to evaluate the efficacy of Dexamethasone and Methylprednisolone as a treatment for severe Acute Respiratory Distress Syndrome (ARDS) caused by coronavirus disease 19 (COVID-19). Our aim is to find the best option for the treatment and management of ARDS in COVID-19 patients.

ELIGIBILITY:
Inclusion Criteria:

• Moderate to severe COVID-19 requires hospitalization. SARS-CoV-2 infection will be confirmed by RT PCR / CT Chest in every case.

Exclusion Criteria:

* Participants with uncontrolled clinical status who were hospitalized from the before.
* Contraindication / possible drug interaction.
* Participants who have any severe and/or uncontrolled medical conditions like, Severe ischemic heart disease, epilepsy, malignancy, Pulmonary/renal/hepatic disease, pregnancy, Corpulmonale, etc.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-08-02 (Actual); Primary Completion 2020-11-15 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
Mortality rate (In hospital) | Following randomization 30 days.
Clinical improvement | Following randomization 30 days.
  The number of participants with "Clinical improvement" determined by the improvement of individual presenting symptoms of the COVID19; changes in radiological and laboratory values.Patient admitted in general bed requiring High Dependency Unit (HDU), and an HDU patient requiring Ventilator or Intensive care support.

SECONDARY OUTCOMES:
Ventilator free days | Following randomization 30 days.
Changes in Oxygen level | Following randomization 30 days.
  Oxygen saturation in the peripheral blood determined by pulse oximetry.

CONTACTS AND LOCATIONS:
Overall Officials: Abu Taiub Mohammed Mohiuddin Chowdhury, MBBS, MD, Study Director — First Affiliated Hospital Xi'an Jiaotong University; Abu Taiub Mohammed Mohiuddin Chowdhury, MBBS, MD, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (2):
- Bangladesh (2):
  - Chattogram General Hospital, Chittagong
  - M. Abdur Rahim Medical College Hospital, Dinajpur

IPD SHARING:
Plan to Share IPD: No